CLINICAL TRIAL: NCT03063853
Title: Early Versus Late Removal of Surgical Staples After Cesarean Delivery. Randomized Control Trial.
Brief Title: Removal of Surgical Staples After Cesarean Delivery. Randomized Control Trial.
Acronym: ROCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0150-16- WOMC
Record Dates: First submitted 2017-02-22; First posted 2017-02-24 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-02

CONDITIONS: Cesarean Section; Wound, Infection (Following Delivery)
MeSH Terms: conditions — Wounds and Injuries; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POD4 (Other): REMOVAL OF SURGICAL STAPLES AT POSTOPERATIVE DAY 4
  Interventions: Other: Removal of surgical clips at day 4 post operative vs day 8 post operative; Procedure: Elective cesarean delivery
- POD8 (Other): REMOVAL OF SURGICAL STAPLES AT POSTOPERATIVE DAY 8
  Interventions: Other: Removal of surgical clips at day 4 post operative vs day 8 post operative; Procedure: Elective cesarean delivery

INTERVENTIONS:
Other: Removal of surgical clips at day 4 post operative vs day 8 post operative — Removal of surgical clips at day 4 post operative vs day 8 post operative
Procedure: Elective cesarean delivery — non emergent elective cesarean delivery

SUMMARY:
The optimal choice of skin closure at cesarean delivery has not yet been determined. This study aim to study the wound complications and scar healing after Surgical staples removal at postoperative day 4 and day 8 .

A randomized control trial.

DETAILED DESCRIPTION:
A randomized controlled trial in which pregnant women undergoing a scheduled Elective cesarean delivery were assigned to skin closure with surgical staples and were randomly assigned to the day of removal of surgical staples. Postoperative day 4 VS. Postoperative day 8 .

Outcome assessors were blinded to group allocation. Scars will be evaluated after 8 weeks. Primary outcome measures is Patient and Observer Scar Assessment Scale (POSAS) scores. Secondary outcome measures are complications of surgical site infection (SSI) or wound disruption (hematoma or seroma).

A group of 104 women is needed in order to achieve a clinically signiﬁcant effect with a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean delivery
* previous cesarean delivery performed using the Pfannenstiel method
* 36-41 weeks of gestation based on first trimester ultrasound and a viable fetus.

Exclusion Criteria:

* emergency cesarean delivery
* clinical signs of infection at the time of CD, uncontrolled
* vunblanaced diabetes mellitus
* history of keloids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) scores. | 8 weeks postoperative

SECONDARY OUTCOMES:
complications of surgical site infection (SSI) or wound disruption (hematoma or seroma). | 8 weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Miremberg, MD, Principal Investigator — Wolfson Medical Center- Tel Aviv University
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: No